CLINICAL TRIAL: NCT04948814
Title: Clinical Trial of Fecal Microbiota Transplantation in Children With Autism Spectrum Disorder
Brief Title: Application of Fecal Microbiota Transplantation in Children With ASD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Yan Hao, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F616
Record Dates: First submitted 2021-06-21; First posted 2021-07-02 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder，Fecal microbiota transplantation
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Fecal Microbiota Transplantation; Vancomycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASD children (Experimental): 20 ASD children who meet the eligibility requirements will receive a fecal microbiota transplantation following a 2-week treatment with Vancomycin (40mg/kg/day) after 3 month waiting period. Fresh stool sample will be obtained from the donor. Fecal bacteria transplantation will be achieved via endoscopy, nasogastric/nasointestinal tubes, the proximal colon by colonoscopy, or the distal colon by enema, rectal tube, or sigmoidoscopy or a combined approach. The amount of fecal bacterial liquid transplantation for children is 5ml/kg each time. Fecal microbiota transplantation will be conducted at week 3-4, week 6-7, week 9, week 11 and week 13 for total 5 round.
  Interventions: Biological: Fecal microbiota transplantation; Drug: Vancomycin

INTERVENTIONS:
Biological: Fecal microbiota transplantation — FMT utilizing stool from healthy children
Drug: Vancomycin — 40mg/kg/day

SUMMARY:
Autism Spectrum Disorder (ASD) is a group of serious neurodevelopmental disorders. Intestinal microbial disturbance is common in children with ASD, and about 40% of ASD children suffer from gastrointestinal dysfunction. A great deal of evidence shows that intestinal microbes can influence the brain to play its role through "brain-intestinal-microbiota axis". Fecal microbial biota transplantation (FMT) is the most direct way to change the intestinal flora rapidly. We intend to study the difference of intestinal flora structure and metabolism between ASD children and control children at the level of phylum, genus and species; To explore the role of fecal bacteria transplantation in improving core symptoms and gastrointestinal dysfunction of children in autism spectrum disorder; To study the potential etiological mechanism of autism spectrum disorder.

DETAILED DESCRIPTION:
20 ASD children and 20 healthy children who are 3 to 18 years of age will be enrolled in the trial. The fecal donors who are 20 healthy children, will be extensively screened for infectious diseases prior to providing stool for the transplant. After being informed about the study and potential risks, all patients giving written informed consent will undergo screening period to determine eligibility for study entry. 20 ASD children who meet the eligibility requirements will receive a fecal microbiota transplantation following a 2-week treatment with Vancomycin. Fecal bacteria transplantation will be achieved through nasogastric tube, nasojejunal tube, esophagogastroduodenoscopy, colonoscopy or enema. The amount of fecal bacterial liquid transplantation for children is 5ml/kg each time. Microbiota analysis will also be performed on both the donor and recipient stool sample prior to transplantation, and on the recipient sample at 1 month, 3 month and 6 months post transplantation. We evaluate the difference of intestinal flora structure and metabolism between ASD children and control children at the level of phylum, genus and species, and explore the role of fecal bacteria transplantation in improving core symptoms and gastrointestinal dysfunction of children in autism spectrum disorder.

ELIGIBILITY:
Inclusion criteria for ASD children.

1. Children who meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) and ADOS-2 diagnostic criteria.
2. Age 3-18 years.

Inclusion criteria for donor.

1. Children who match ASD children in age and gender, preferably from relatives.
2. No antibiotic treatment in the last 3 months.
3. Children who are healthy in growth and development, with normal results of child developmental and neuropsychological tests, including ASD-related screening, Attention-deficit hyperactivity disorder (ADHD)-related screening and motor screening.
4. Children who have normal serological test results, including pre-transfusion testing, liver and kidney function, hepatitis B detection, quantification of hepatitis C, quantification of A virus immunoglobulin M (HAV-IgM), Epstein-Barr virus DNA (EBV-DNA) and Human Immunodeficiency Virus (HIV), detection of microvirus B19, TORCH, tuberculosis infection T-cell test (T-SPOT), total total immunoglobulin E (IgE), food and inhalant allergen testing, and lymphocyte subpopulation analysis.
5. Children who have normal stool test results, including fecal routine and fecal occult blood, bacteria (Clostridium difficile A/B toxin, Escherichia coli O157, Shigella spp., Salmonella spp., Campylobacter spp., Staphylococcus aureus, Yersinia spp., Vibrio parahaemolyticus, Cholera isolates), fungi (Pseudomonas albicans, etc.), viruses (rotavirus, etc.), parasites (Giardia lamblia, Cryptosporidium, Cyclospora).
6. Children who have normal results for chest X-ray, abdominal ultrasound, C13 breath test, cranial MRI, etc.

Exclusion criteria for ASD children.

1. ASD children with severe gastrointestinal symptoms or organic disease requiring immediate surgery or treatment.
2. ASD children who have received antibiotics within 3 months, or are receiving immunosuppressive agents and biologics.
3. ASD children with underlying diseases, such as severe anemia, malnutrition, autoimmune diseases (autoimmune thyroiditis, type I diabetes, etc.), allergic diseases (asthma, severe eczema, etc.), central nervous system diseases, metabolic syndrome, etc.
4. ASD children with other organic dysfunctions, such as cerebral palsy, congenital genetic diseases, etc.; history of other psychiatric-behavioral disorders, genetic-metabolic diseases and other major physical diseases; other physical diseases, such as hearing impairment, vocal disorders, blindness, etc.

Exclusion criteria for donor.

1. Children who have functional gastrointestinal symptoms suggested by the Rome IV diagnostic questionnaire for functional gastrointestinal disorders.
2. Children who have gastrointestinal disorders, including gastrointestinal symptoms (e.g., nausea, vomiting, abdominal pain, bloating, diarrhea, constipation, etc.), chronic gastrointestinal disorders (chronic diarrhea, chronic abdominal pain, etc.), gastroesophageal reflux disease, peptic ulcer, a history of gastrointestinal surgery (intestinal obstruction, megacolon, pyloric stenosis, etc.)
3. Children who suffer from other diseases, including familial autoimmune diseases such as type I diabetes, inflammatory bowel disease, rheumatoid arthritis, chronic lymphocytic thyroiditis (Hashimoto's disease), toxic diffuse goiter (Graves' disease), etc.;
4. Children who have received drugs that has impact on the intestinal microbiota (such as proton pump inhibitors, pro-gastrointestinal drugs, steroids, aspirin, etc.) within six months.
5. Children who have received antibiotics within three months;
6. Children who are receiving immunosuppressants and biological agents.
7. Children who are undergoing chemotherapy for various tumors;
8. Children who have liver and kidney diseases, central nervous system diseases, acute and chronic infectious diseases (tuberculosis, measles, syphilis, HIV, etc.), severely anemic, malnourished, metabolic syndrome (obesity, diabetes, etc.),
9. Children who live in a place with prevalence of bacterial, viral, parasitic, etc.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Autism Diagnostic Observation Scale (ADOS) in ASD children | baseline, 2 weeks, 5 weeks , 8 weeks , 10 weeks , 12 weeks and 14 weeks, and 1 month, 3 month, 6 months post transplantation
  The ADOS consists of a series of structured and semi-structured tasks that involve social interaction between the examiner and the person under assessment. The examiner observes and identifies segments of the subject's behavior and assigns these to predetermined observational categories. Categorized observations are subsequently combined to produce quantitative scores for analysis and diagnostic classification of ASD. Children at or above predetermined cutoff lines are considered to be positive for ASD. The assessment will be conducted before and after each intervention, namely baseline, 2 weeks, 5 weeks , 8 weeks , 10 weeks , 12 weeks and 14 weeks, and 1 month, 3 month, 6 months post transplantation.
Changes in the Autism Behavior Checklist (ABC) in ASD children | baseline, 2 weeks, 5 weeks , 8 weeks , 10 weeks , 12 weeks and 14 weeks, and 1 month, 3 month, 6 months post transplantation
  ABC is a scale used for nonadaptive behaviors created to screen and indicate the probability of a diagnosis of autism. The questionnaire including 57 items related to five areas: sensorial, relational, use of body and objects, and social skills. Scale score> 67 strongly suggests the presence of autism. The assessment will be conducted before and after each intervention, namely baseline, 2 weeks, 5 weeks , 8 weeks , 10 weeks , 12 weeks and 14 weeks, and 1 month, 3 month, 6 months post transplantation.
Changes in the Childhood Autism Rating Scale (CARS) in ASD children | baseline, 2 weeks, 5 weeks , 8 weeks , 10 weeks , 12 weeks and 14 weeks, and 1 month, 3 month, 6 months post transplantation
  CARS assesses the child on a scale from 1 to 4 in each of 15 dimensions or symptoms. A total score of at least 30 strongly suggests the presence of autism. Children with score between 30 and 36 have mild-to-moderate autism while those with score between 37 and 60 have severe autism. The assessment will be conducted before and after each intervention, namely baseline, 2 weeks, 5 weeks , 8 weeks , 10 weeks , 12 weeks and 14 weeks, and 1 month, 3 month, 6 months post transplantation.
Change in Social Responsiveness Scale (SRS) in ASD children | baseline, 2 weeks, 5 weeks , 8 weeks , 10 weeks , 12 weeks and 14 weeks, and 1 month, 3 month, 6 months post transplantation
  The SRS is a 65-item rating scale with standardized measure of the core symptoms of autism. Each item is scored on a 4-point Likert scale. The score of each individual item is summed to create a total raw score. A total scores results are as follows:
  0-62: Within normal limits 63-79: Mild range of impairment 80-108: Moderate range of impairment 109-149: Severe range of impairment. The assessment will be conducted before and after each intervention, namely baseline, 2 weeks, 5 weeks , 8 weeks , 10 weeks , 12 weeks and 14 weeks, and 1 month, 3 month, 6 months post transplantation.
Change in Autism Treatment Evaluation Checklist (ATEC) in ASD children | baseline, 2 weeks, 5 weeks , 8 weeks , 10 weeks , 12 weeks and 14 weeks, and 1 month, 3 month, 6 months post transplantation
  ASD symptoms will be assessed using the Chinese version of the Autism Treatment Evaluation Checklist (ATEC), which comprise four subscales to measure child speech/language/communication, sociability, sensory/cognitive awareness, and health/physical/behavior. The scale has 77 items that are scored by parents. The health/physical/behavior subscale is rated using a 0 (not a problem)-to-3 (serious problem) point scale, whereas the other three subscales are rated using a 0 (not true)-to-2 (very true) point scale. Higher scores represent more ASD symptoms. The assessment will be conducted before and after each intervention, namely baseline, 2 weeks, 5 weeks , 8 weeks , 10 weeks , 12 weeks and 14 weeks, and 1 month, 3 month, 6 months post transplantation.
Change in gastrointestinal symptoms among children with ASD | baseline, 2 weeks, 5 weeks , 8 weeks , 10 weeks , 12 weeks and 14 weeks, and 1 month, 3 month, 6 months post transplantation
  Assessment will be conducted for the Rome IV diagnoses of cyclic vomiting, functional vomiting, functional dyspepsia, and/or functional constipation. The presence or absence of meeting criteria for the Rome IV diagnoses will be coded as a binary variable (true/false) to represent resolution of symptoms. The assessment will be conducted before and after each intervention, namely baseline, 2 weeks, 5 weeks , 8 weeks , 10 weeks , 12 weeks and 14 weeks, and 1 month, 3 month, 6 months post transplantation.
Evaluate the difference of the gut microbe composition between children with ASD and healthy children by sequencing faecal metagenome. | 6 months post transplantation
  Fecal samples from ASD and healthy children were collected at baseline, 2 weeks, 5 weeks , 8 weeks , 10 weeks , 12 weeks and 14 weeks, and 1 month, 3 month, 6 months post transplantation.The composition of the gut microbe was evaluated by sequencing faecal metagenome. We evaluate the differences in the structure of the flora and its metabolism between the two at the phylum, genus and species levels of the intestinal flora and control children, and to develop a model for predicting the structure of the flora.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Background] Fattorusso A, Di Genova L, Dell'Isola GB, Mencaroni E, Esposito S. Autism Spectrum Disorders and the Gut Microbiota. Nutrients. 2019 Feb 28;11(3):521. doi: 10.3390/nu11030521. PMID 30823414
- [Background] Israelyan N, Margolis KG. Serotonin as a link between the gut-brain-microbiome axis in autism spectrum disorders. Pharmacol Res. 2018 Jun;132:1-6. doi: 10.1016/j.phrs.2018.03.020. Epub 2018 Mar 31. PMID 29614380
- [Background] Fetissov SO, Averina OV, Danilenko VN. Neuropeptides in the microbiota-brain axis and feeding behavior in autism spectrum disorder. Nutrition. 2019 May;61:43-48. doi: 10.1016/j.nut.2018.10.030. Epub 2018 Oct 27. PMID 30684851
- [Background] Mussap M, Noto A, Fanos V. Metabolomics of autism spectrum disorders: early insights regarding mammalian-microbial cometabolites. Expert Rev Mol Diagn. 2016 Aug;16(8):869-81. doi: 10.1080/14737159.2016.1202765. Epub 2016 Jun 30. PMID 27310602
- [Background] Adams JB, Audhya T, McDonough-Means S, Rubin RA, Quig D, Geis E, Gehn E, Loresto M, Mitchell J, Atwood S, Barnhouse S, Lee W. Nutritional and metabolic status of children with autism vs. neurotypical children, and the association with autism severity. Nutr Metab (Lond). 2011 Jun 8;8(1):34. doi: 10.1186/1743-7075-8-34. PMID 21651783